CLINICAL TRIAL: NCT02463617
Title: Impulsivity and Parkinson's Disease : a Neuropsychology With Magnetic Resonance Imaging Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IMPULSPARK
Record Dates: First submitted 2015-02-13; First posted 2015-06-04 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PD patients (Other)
  Interventions: Other: magnetic resonance imaging

INTERVENTIONS:
Other: magnetic resonance imaging

SUMMARY:
This study aims to characterize the nature of impulsivity in Parkinson's Disease (PD).

ELIGIBILITY:
Inclusion criteria :

Early onset PD patients and late onset PD patients with siblings available PD patients with or without impulse control disorders Current or past treatment with dopamine agonists or levodopa PD patients without dementia Age < 80 ans

Exclusion criteria :

Early onset PD patients and late onset PD patients without siblings available PD patients with dementia Age > 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-11-21 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Barratt Impulsiveness Scale | up to three months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc HOUETO, MD PhD, Principal Investigator — Poitiers University Hospital, France
Locations (3):
- France (3):
  - Pascal DERKINDEREN, Nantes
  - Chu de Poitiers, Poitiers
  - Marc VERIN, Rennes